CLINICAL TRIAL: NCT01898481
Title: Triadic Expectations: Decision Making in the Context of Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00045101
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Health Care Decision Making
Keywords: Health care decision making

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health Care Triads: This is an exploratory pilot study of 25 health care triads. Triads will include: (1) a patient diagnosed with advanced cancer, (2) a loved one, and (3) an oncology provider.

SUMMARY:
The purpose of this pilot study is to test the feasibility of identifying and interviewing healthcare triads (patients, loved ones and oncologists) in a research study and evaluate the influences of patients' loved ones and oncologists on cancer treatment decision-making. the study team plans to explore concordance or discordance within the triad about the decisions, and also assess decisional conflict, regret and distress. Study methods involve interviewing a total of 75 patients, their loved ones and oncologists about past cancer treatment decisions. Analysis will consist mainly of qualitative content analysis. The investigators do not anticipate risk or safety issues beyond loss of confidentiality or minimal discomfort while discussing a cancer treatment decision.

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate the influences of oncologists and patients' loved ones on cancer treatment decision-making. The specific aims are:

AIM 1: Test the feasibility of identifying and interviewing health care triads (patients, loved ones, and oncologists) in a research study about treatment decisions.

AIM 2: Assess perceptions of the decision-making experience from the perspective of three parties within the health care triad (patients, loved ones, and oncologists) and examine the relationships among the triadic perspectives.

AIM 3: Explore concordance or discordance within the triad about cancer treatment decisions and assess decisional conflict, decisional regret, and distress.

This is an exploratory pilot study of 25 health care triads. Triads will include: (1) a patient diagnosed with advanced cancer, (2) a loved one, and (3) an oncology provider. In a few instances, the study team may interview more than one oncologist or loved one per patient.

In phase one of recruitment, oncologists will be recruited and enrolled. In phase two, the study team will recruit patients who receive care from at least one enrolled oncologist and at least one of the patient's friends or family members. While oncology providers may participate in the study with multiple patients and their loved ones, the patients will be unique to each triad.

Investigators anticipate enrolling two triads per week for a total of three months. They will utilize mainly qualitative methods, and specifically, content analysis, in this exploratory pilot study to (1) further hone and develop research questions and aims for a larger study with appropriate statistical power, (2) test the feasibility of recruiting health care triads in the oncology context, and (3) strengthen our study design, protocols and surveys. The investigators plan to use an iterative process of coding to allow for protocol and survey revisions, and in particular the inclusion of new probes, during the study. The codebook will include inductive and deductive codes related to the general decision making process, expectations and decisional outcomes, conflict and concordance between members of the triad, and other relevant topics. Two coders will review each interview and the team will review for themes and exemplars. The investigators plan to pilot three scales in this study that might be used in a larger future study.

ELIGIBILITY:
Oncologist Inclusion Criteria:

* At least 18 years of age;
* An attending physician or fellow at Duke University Medical Center;
* Medical, surgical or radiation oncologist;
* Provides care to patients diagnosed with at least one of the following conditions:

  * Recurrent or refractory Acute Myeloid Leukemia (AML), also known as acute myelogenous leukemia or acute nonlymphocytic leukemia (ANLL);
  * Chronic myeloid leukemia (CML) in blast phase;
  * Non-hodgkin lymphoma (NHL), relapsed or refractory;
  * Acute lymphocytic leukemia (ALL), relapsed or refractory;
  * Metastatic pancreatic cancer;
  * Metastatic colorectal cancer;
  * Metastatic gastro-esophageal cancer;
  * Metastatic Cholangiocarcinoma.

Patient Inclusion Criteria:

* At least 18 years of age;
* A Duke patient receiving care from an oncology provider who is enrolled in the study;
* Currently admitted to the Duke University hematological malignancies in-patient service OR being seen at Duke's outpatient GI cancer clinic;
* Made a cancer treatment decision in the last 3 months;
* Diagnosed with one of the following:

  * Recurrent or refractory Acute Myeloid Leukemia (AML), also known as acute myelogenous leukemia or acute nonlymphocytic leukemia (ANLL);
  * Chronic myeloid leukemia (CML) in blast phase;
  * Non-hodgkin lymphoma (NHL), relapsed or refractory;
  * Acute lymphocytic leukemia (ALL), relapsed or refractory;
  * Metastatic pancreatic cancer;
  * Metastatic colorectal cancer;
  * Metastatic gastro-esophageal cancer;
  * Metastatic Cholangiocarcinoma.

Loved One (friend/family) Inclusion Criteria:

* At least 18 years of age;
* Identified by patient as influential in a recent (within 3 months) treatment decision;
* Able and willing to complete the study interview in person or by telephone.

Exclusion for all Subjects:

* Lacking capacity to give legally effective consent;
* Does not read or understand English.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer, their friends/family, and oncologists
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Decisional Regret | three to four months after treatment decision
  This outcome will be measured with an interviewer-administered survey.
Decisional concordance or discordance among members of triads | three to four months after treatment decision
  This outcome will be measured with an interviewer-administered survey.

CONTACTS AND LOCATIONS:
Overall Officials: James Tulsky, MD, Principal Investigator — Duke University; Dan Ariely, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States